CLINICAL TRIAL: NCT02318381
Title: Suprascapular Neuropathy in the Setting of Rotator Cuff Tears; Results of Arthroscopic Treatment
Brief Title: Suprascapular Neuropathy in the Setting of Rotator Cuff Tears: Results of Arthroscopic Treatment
Acronym: SupraCufTear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Nikolaos Platon Sachinis, Dr Nikolaos Platon Sachinis, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSachinisPhD1
Record Dates: First submitted 2014-12-05; First posted 2014-12-17 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Entrapment Neuropathy; Rotator Cuff Tear
Keywords: suprascapular nerve; rotator cuff tear; suprascapular neuropathy; superior transverse scapular ligament
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients with suprascapular neuropathy and rotator cuff tear treated arthroscopically without release of the superior transverse scapular ligament.
- Ligament Release (Other): Patients with suprascapular neuropathy and rotator cuff tear treated arthroscopically with release of the suprascapular nerve.
  Arthroscopic dissection of the superior transverse scapular ligament
  Interventions: Procedure: Dissection of the superior transverse scapular ligament

INTERVENTIONS:
Procedure: Dissection of the superior transverse scapular ligament — After treatment of the rotator cuff tear, the arthroscopic procedure will also proceed with the dissection of the superior transverse scapular ligament, in order to release pressure from the suprascapular nerve.
  Arms: Ligament Release

SUMMARY:
Aim of this prospective double blind randomized clinical trial is to understand the correlation of suprascapular neuropathy in the setting of large and massive tears of the shoulder rotator cuff and to investigate whether arthroscopic dissection of the superior transverse scapular ligament is positively related to the improvement of this neuropathy.

DETAILED DESCRIPTION:
The suprascapular nerve originates from the upper trunk of the brachial plexus with participation from the A5 and A6 spinal nerve roots and occasionally from the A4 root. It is treading behind the clavicle and to the upper border of the scapula and then enters through the scapular notch of the shoulder and below the transverse superior transverse ligament to the rear surface of the scapula. This entry point is an important factor of pressure and surgical dissection of the ligament enlarges the space through which the nerve travels.

The rotator cuff consists of the tendons of subscapularis, supraspinatus , infraspinatus and minor teres muscles. Cadaveric studies have shown that tears in the cuff , particularly massive ruptures a gap more than 5cm, change the path of the suprascapular nerve and create conditions that pressure.

Until now, there are no prospective studies that compare the improvement of suprascapular neuropathy after arthroscopic dissection of the superior transverse scapular ligament in patients with rotator cuff tears , or that study the degree of neuropathy compared with the extent of the rupture .

ELIGIBILITY:
Inclusion Criteria:

- Large of Massive repairable rotator cuff tears combined suprascapular neuropathy

Exclusion Criteria:

* Suprascapular neuropathy of another cause (eg. brachial plexus neuropathy)
* Other surgery at the same shoulder region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2018-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Changes of function of suprascapular nerve, assessed by electromyographic (EMG) and nerve conduction studies (NCS). | Up to 6 weeks prior to surgery, at 6 months and at one year post-operatively.
  Abnormal function of the suprascapular nerve in EMG studies will be indicated by fibrillation and high- frequency discharge potentials. An abnormal NCS finding is defined according to following values: infraspinatus latency >4.5ms and amplitude <8mV from peak to peak and supraspinatus muscle latency >3.5 ms and an amplitude <8 mV from peak to peak. The contralateral nerve will also be examined. Abnormal findings are also indicated when the difference in amplitude to the healthy side is >50%.

SECONDARY OUTCOMES:
Size of rotator cuff tear | Up to 6 weeks prior to surgery
  Size of rotator cuff tear will be measured in magnetic resonance tomography images, according to Cofield Classification of Rotator Cuff Tears (Cofield, Surg Gynec Obstet, 154(5): 667-672, 1982). Classification follows: Small tear < 1cm, Medium 1-3 cm, Large 3-5 cm, Massive >5cm. Diameter of the tear is measured.
Changes of fatty infiltration of rotator cuff muscles | Up to 6 weeks prior to surgery, one year post-operatively.
  Fatty infiltration is assessed with magnetic resonance imaging studies, according to Goutallier's classification (Goutallier et al, CORR, 304:78-83, 1994). Classification follows: Stage 0 - Normal muscle, Stage 1 - Some fatty streaks, Stage 2 - Less than 50% fatty muscle atrophy, Stage 3 - 50% fatty muscle atrophy, Stage 4 - Greater than 50% fatty muscle atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Sachinis, M.D., Principal Investigator — First Orthopaedic Department of Aristotle University of Thessaloniki; Pericles Papadopoulos, Ph.D., Study Chair — First Orthopaedic Department of Aristotle University of Thessaloniki; Sotirios Papagianopoulos, Ph.D., Study Director — Τhird Neurology Department of Aristotle University of Thessaloniki; Ioannis Sarris, Ph.D., Study Director — Third Orthopaedic Department of Aristotle University of Thessaloniki
Locations (1):
- First Orthopaedic Department of Aristotle University of Thessaloniki, 'G. Papanikolaou' Hospital, Thessaloniki, Exohi, Greece

REFERENCES:
- [Result] Collin P, Treseder T, Ladermann A, Benkalfate T, Mourtada R, Courage O, Favard L. Neuropathy of the suprascapular nerve and massive rotator cuff tears: a prospective electromyographic study. J Shoulder Elbow Surg. 2014 Jan;23(1):28-34. doi: 10.1016/j.jse.2013.07.039. Epub 2013 Sep 30. PMID 24090983
- [Result] Costouros JG, Porramatikul M, Lie DT, Warner JJ. Reversal of suprascapular neuropathy following arthroscopic repair of massive supraspinatus and infraspinatus rotator cuff tears. Arthroscopy. 2007 Nov;23(11):1152-61. doi: 10.1016/j.arthro.2007.06.014. PMID 17986401
- [Result] Lafosse L, Tomasi A, Corbett S, Baier G, Willems K, Gobezie R. Arthroscopic release of suprascapular nerve entrapment at the suprascapular notch: technique and preliminary results. Arthroscopy. 2007 Jan;23(1):34-42. doi: 10.1016/j.arthro.2006.10.003. PMID 17210425
- [Result] Albritton MJ, Graham RD, Richards RS 2nd, Basamania CJ. An anatomic study of the effects on the suprascapular nerve due to retraction of the supraspinatus muscle after a rotator cuff tear. J Shoulder Elbow Surg. 2003 Sep-Oct;12(5):497-500. doi: 10.1016/s1058-2746(03)00182-4. PMID 14564276
- [Result] Greiner A, Golser K, Wambacher M, Kralinger F, Sperner G. The course of the suprascapular nerve in the supraspinatus fossa and its vulnerability in muscle advancement. J Shoulder Elbow Surg. 2003 May-Jun;12(3):256-9. doi: 10.1016/s1058-2746(02)00034-4. PMID 12851579
- [Derived] Sachinis NP, Papagiannopoulos S, Sarris I, Papadopoulos P. Outcomes of Arthroscopic Nerve Release in Patients Treated for Large or Massive Rotator Cuff Tears and Associated Suprascapular Neuropathy: A Prospective, Randomized, Double-Blinded Clinical Trial. Am J Sports Med. 2021 Jul;49(9):2301-2308. doi: 10.1177/03635465211021834. Epub 2021 Jun 22. PMID 34156877
- [Derived] Sachinis NP, Boutsiadis A, Papagiannopoulos S, Ditsios K, Christodoulou A, Papadopoulos P. Suprascapular neuropathy in the setting of rotator cuff tears: study protocol for a double-blinded randomized controlled trial. Trials. 2016 Nov 22;17(1):554. doi: 10.1186/s13063-016-1672-y. PMID 27876086